CLINICAL TRIAL: NCT05576727
Title: Prediction of Development and Rupture Risk for Intracranial Unruptured Aneurysms
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Jinhua Central Hospital (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); The Central Hospital of Lishui City (Other); Ningbo Medical Center Lihuili Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: UNruAneu
Record Dates: First submitted 2022-10-10; First posted 2022-10-12 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Unruptured Intracranial Aneurysm
  Interventions: Other: Unruptured intracranial aneurysms

INTERVENTIONS:
Other: Unruptured intracranial aneurysms — Extensive clinical, biological and imaging data of unruptured intracranial aneurysm patients will be recorded during a 5 years follow-up.

SUMMARY:
In recent years, researches on the natural history and risk factors of intracranial unruptured aneurysms have become a hot topic at home and abroad. However, risk factors for aneurysm rupture is still unclear yet. The investigators' preliminary study focused on constructing a rupture risk prediction system for intracranial unruptured aneurysm in the investigators' single center. The investigators' result showed that three significant factors (sex, abnormal serum tumor necrosis factor (TNF)-α and coincidence of thin-walled regions (TWR) and normalized wall shear stress (NWSS)) stood out by using logistic regression to explore the rupture risk factors of intracranial unruptured aneurysms, which could help guide the clinical treatment of intracranial unruptured aneurysms. This study is to evaluate and improve the rupture predict model of intracranial unruptured aneurysm in multi-neurosurgical centers.

DETAILED DESCRIPTION:
In recent years, researches on the natural history and risk factors of intracranial unruptured aneurysms have become a hot topic at home and abroad. However, risk factors for aneurysm rupture is still unclear yet. The investigators' preliminary study focused on constructing a rupture risk prediction system for intracranial unruptured aneurysm in the investigators' single center. Four aspects for unruptured aneurysms were collected: (1) Patients' basic demographic characteristics; (2) Reconstruction of intracranial unruptured aneurysm wall with 7-Tesla MRI, and explore the technical parameters of 7-Tesla high-resolution black blood MRI scanning intracranial aneurysm wall (0.5 mm isotropic resolution), as well as assessing the relationship between aneurysm wall enhancement (AWE), thin-walled regions (TWR), and hemodynamic parameters and their relationship to aneurysm development; (3) Using hydrodynamics to explore the hemodynamic parameters of intracranial unruptured aneurysms, explore new hydrodynamic parameters and screen rupture-related risk factors; (4) The use of single-cell RNA sequencing technology to explore the infiltration of immune cells in the aneurysm wall tissue of intracranial unruptured aneurysms. Based on the above research results, three significant factors (sex, abnormal serum TNF-α and coincidence of TWR and normalized wall shear stress (NWSS)) stood out by using logistic regression to explore the rupture risk factors of intracranial unruptured aneurysms, which could help guide the clinical treatment of intracranial unruptured aneurysms. This study is to evaluate and improve the rupture predict model of intracranial unruptured aneurysm in multi-neurosurgical centers.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of aneurysm by digital subtraction angiography (DSA);
2. Age between 18-70 years old;
3. Informed consent form for this study was signed

Exclusion Criteria:

1. Dissecting aneurysms and saccular aneurysms with other vascular diseases such as arteriovenous malformations, moyamoya disease, and arteriovenous fistulas were excluded;
2. Combined with serious systemic diseases;
3. Patients who cannot receive MRI/magnetic resonance angiography (MRA) examinations due to severely impaired renal function, allergy, space claustrophobia or internal implants in the body.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The enrolled patients are who have unruptured asymptomatic aneurysm with a clinical, a biological and an imaging follow-up, without any relative treatment.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Predictive value of coincidence of TWR and NWSS for unruptured aneurysm rupture | at 5 year
  at 5 years, the value of the factor (coincidence of TWR and NWSS) to predict aneurysm rupture risk will be analyzed
Predictive value of serum TNF-α for unruptured aneurysm rupture | at 5 year
  at 5 years, the value of the factor (serum TNF-α) to predict aneurysm rupture risk will be analyzed
Predictive value of sex for unruptured aneurysm rupture | at 5 year
  at 5 years, the value of the factor (sex) to predict aneurysm rupture risk will be analyzed

SECONDARY OUTCOMES:
Predictive value of coincidence of TWR and NWSS for unruptured aneurysm growth | at 5 year
  at 5 years, the value of the factor (coincidence of TWR and NWSS) to predict aneurysm growth risk will be analyzed
Predictive value of serum TNF-α for unruptured aneurysm growth | at 5 year
  at 5 years, the value of the factor (serum TNF-α) to predict aneurysm growth risk will be analyzed
Predictive value of sex for unruptured aneurysm growth | at 5 year
  at 5 years, the value of the factor (sex) to predict aneurysm growth risk will be analyzed

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China